CLINICAL TRIAL: NCT07229508
Title: Trajectories of Reinforcement, Activity, and Consumption in Kids
Brief Title: Developmental Trajectories of Reinforcer Pathology and Childhood Obesity
Acronym: TRACK
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00008702; 1R01DK139258-01A1 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Obesity
Keywords: Reinforcer Pathology Theory; Reinforcing Value; Delay Discounting
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aged 8.5-9: Children that are enrolled when they are 8.5- 9 years, 11 months of age
- Aged 10.5-11: Children that are enrolled when they are 10.5-11 years, 11 months age

SUMMARY:
The goal of this observational study is to understand how children's food preferences, physical activity, and decision-making change over time and how these behaviors relate to body weight and overall health.

DETAILED DESCRIPTION:
A cohort sequential design will be used to track 2 cohorts of children aged 8.5-9 years 11 months, and 10.5-11 years 11 months over a 3 year period to understand how the development of food and activity reinforcement and delay discounting could lead to the development of childhood obesity in children aged 9-14.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children
* Black, Indigenous, and People of Color (BIPOC) or Hispanic families
* Children from low SES families (as defined by household education, eligibility for government assistance)
* Children in overweight/obese category (defined by range in each cohort)

Exclusion Criteria:

* Medical causes for obesity
* Stature below the 5th percentile
* Physical activity restrictions
* Psychopathology
* Medication use that affects activity or appetite
* Children that spend less than 65% of their time in participating parent's household
* BMI percentile criteria
* Liking of study foods and activities
* Dietary restrictions and food allergies

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male and female children of varying racial/ethnic backgrounds, SES backgrounds, and varying body compositions
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
zBMI | 0, 12, 24 and 36 months
  Height and weight will be measured to determine zBMI using the CDC extended BMI-for-age growth charts. First, height (m) and weight (kg) will be used to calculate BMI (kg/m^2), then, using the CDC extended BMI-for-age growth charts, a zBMI score will be determined based on the charts.
body fat | 0, 12, 24 and 36 months
  Body fat (% of body weight) will be measured using the Tanita BF-400 Total Body Analyzer.
percent change over the overweight BMI | 0, 12, 24 and 36 months
  Height and weight will be measured to calculate changes in overweight status of children. Change in percent overweight from 0, 12, 24, 36 months. First, height and weight will be used to calculate BMI (kg/m^2), then CDC extended growth charts will be used to determine BMI percentile. Percent overweight is calculated as ((childBMI percentile - 85th BMI percentile)/(85th BMI percentile)) x 100. Percent over the age- and sex- specific 85th BMI percentile for children will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Epstein, PhD, Principal Investigator — SUNY-University at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No